CLINICAL TRIAL: NCT04620525
Title: The Link Between Cognitive Function and Chronic Pain: An Observational Cohort Study
Brief Title: Cognition, Pain and Wellbeing
Acronym: CPW
Status: Terminated | Type: Observational
Why Stopped: Covid-19 pandemic
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Ana Valdes, Associate Professor, University of Nottingham
Other Study IDs: 1
Record Dates: First submitted 2020-04-22; First posted 2020-11-09 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis
Keywords: knee; osteoarthritis; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood (20ml), urine and faecal samples will be retained to identify inflammatory biomarkers, biomarkers of insulin resistance and gut microbiome measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with the relevant condition: Participants with the relevant condition
- Healthy controls: Healthy controls

SUMMARY:
Osteoarthritis (OA) is the most common form of arthritis and for 4 in 10 people pain from OA is not adequately controlled. The pain experience of people suffering from chronic pain largely depends on their individual perception of pain and on brain functions, in particular what is called "cognitive" functions. Cognitive functions include memory, attention, organisation and planning, task initiation, regulation of emotions and reflection of oneself and are important for everyday tasks, such as following a conversation or a story in a book or on TV, learning new things, remembering old and new information and making decisions. Good cognition predicts the risk of developing chronic pain after a painful event, such as surgery. Chronic pain patients report numerous cognitive impairments, with attention and memory being the two most prominent that can persist even after the original cause of pain has been treated. Little evidence exists regarding the nature and magnitude of these deficits and their underlying brain and psychological mechanisms in chronic knee OA. The investigators want to understand which cognitive functions and to what extent are associated with pain in patients with knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis and for 4 in 10 people pain from OA is not adequately controlled. The pain experience of people suffering from chronic pain largely depends on their individual perception of pain and on brain functions, in particular what is called "cognitive" functions. Cognitive functions include memory, attention, organisation and planning, task initiation, regulation of emotions and reflection of oneself and are important for everyday tasks, such as following a conversation or a story in a book or on TV, learning new things, remembering old and new information and making decisions. Good cognition predicts the risk of developing chronic pain after a painful event, such as surgery. Chronic pain patients report numerous cognitive impairments, with attention and memory being the two most prominent that can persist even after the original cause of pain has been treated. Little evidence exists regarding the nature and magnitude of these deficits and their underlying brain and psychological mechanisms in chronic knee OA. The investigators want to understand which cognitive functions and to what extent are associated with pain in patients with knee OA. Identifying specific domains of cognitive function affected by chronic pain has a clinical utility; specific domains regulate certain aspects of activities of daily living, such as managing personal finances, grocery shopping, remembering to take medications and, thus, dealing with pain early in the disease course could prevent subsequent cognitive loss and long-term pain. To do this the investigators will examine the link between measures of pain and measures of cognition in people with knee OA. The investigators propose to measure knee pain, physical function, sleep quality and overall wellbeing with questionnaires and pain sensitivity measures. The investigators will measure cognition with questionnaires and computer-based tasks testing aspects of cognitive function, including memory and attention. The investigators will compare the questionnaire and pain sensitivity measures with questionnaire and measures of cognitive function in the same participants. The investigators will include tests of various aspects of a person's memory that will facilitate the establishment of which aspects are related to chronic pain. The investigators hypothesise that chronic pain is linked to specific cognitive deficits in patients with knee OA and managing pain, for example, with mild to moderate targeted exercise and healthy diet, may limit the risk of memory loss and dementia and, in turn, predict better treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years and onward
* Able to read and write English
* Have English as their first language

Exclusion Criteria:

* Persons who do not adequately understand verbal explanations of written information in English, or who have special communication needs or whose English is not their first language
* Dialysis patients or on home oxygen
* Terminal illness
* Serious mental illness
* Dementia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from previous studies undertaken by the Academic Rheumatology, University of Nottingham, who have expressed an interest in future research. Responders from the Investigating Musculoskeletal Health and Wellbeing cohort study (IMHWCS, n ~ 5,000) and Knee Pain and related health In the Community cohort study (KPIC, n ~ 3,000) will be sent an invitation letter and participant information sheet (PIS) with details about the Cognition, Pain and Wellbeing study. A telephone screening will be then done to confirm their eligibility for the study and their interest in participating and they will be booked an appointment for a single visit in Academic Rheumatology.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity measures | Conducted once, at assessment visit approximately 10 minutes
  Quantitative sensory testing (QST) will be used to assess pain sensitivity with measures, such as pressure pain threshold (PPT). PPT is a valid measure of tenderness around the knee. QST is used to quantify pain perception and it is an objective measure of peripheral sensitisation (increased tenderness around the knee) and central sensitisation (increased pain perception in areas away from the knee). QST will be used to identify different pain phenotypes among participants and it will enable us to quantify peripheral and central sensitisation components of pain. Pain phenotypes will be then correlated to cognitive measures.
Pain sensitivity measures | Conducted once, at assessment visit approximately 4 minutes
  Quantitative sensory testing (QST) will be used to assess pain sensitivity with measures, such as temporal summation (TS), TS is a measure of central sensitization. QST is used to quantify pain perception and it is an objective measure of peripheral sensitisation (increased tenderness around the knee) and central sensitisation (increased pain perception in areas away from the knee). QST will be used to identify different pain phenotypes among participants and it will enable us to quantify peripheral and central sensitisation components of pain. Pain phenotypes will be then correlated to cognitive measures.
Pain sensitivity measures | Conducted once, at assessment visit approximately 6 minutes
  Quantitative sensory testing (QST) will be used to assess pain sensitivity with measures, such as conditioned pain modulation (CPM). CPM assesses the function of endogenous pain inhibitory pathways. QST is used to quantify pain perception and it is an objective measure of peripheral sensitisation (increased tenderness around the knee) and central sensitisation (increased pain perception in areas away from the knee). QST will be used to identify different pain phenotypes among participants and it will enable us to quantify peripheral and central sensitisation components of pain. Pain phenotypes will be then correlated to cognitive measures.
Pain severity measure | Conducted once, at assessment visit : approximately 5-10 minutes
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), which is a self-administered 24 items questionnaire with three subscales assessing pain, stiffness and physical function, is an extensively utilised tool for the evaluation of hip and knee OA and will be used in the current study.
Cognitive function | Conducted once, at assessment visit : approximately 40 minutes
  Cambridge Neuropsychological Test Automated Battery (CANTAB) (objective measure) including tests of prefrontal-dependent sustained visual attention (Rapid Visual Information Processing, RVP, 7 min), attentional set shifting (Intra-/ Extra- Dimensional Set Shift, IED, 7 min) and hippocampus-dependent paired associate learning (Visual Learning Paired Associates Learning, PAL, 8 min) will be used. Other CANTAB tests will be included for comparison (reaction time test, RTI, 3 min; Stroop-like test, MTT, 8 min; spatial working memory test, SWM, 4 min).
Cognitive function | Conducted once, at assessment visit approximately 8 minutes
  Questionnaire cognitive measures, including the Cognitive Failures Questionnaire (CFQ) will be used.
Cognitive function | Conducted once, at assessment visit approximately 7 minutes
  Questionnaire cognitive measures including the Cognitive reflection test (CRT) will be used.
Neuropathic pain quality: PD-Q | Conducted once, at assessment visit : approximately 5-10 minutes
  The PainDETECT Questionnaire (PD-Q) is a self-report questionnaire developed to discriminate between nociceptive and neuropathic pain. It has been further modified (mPDQ) for use among specific pain groups, for example, knee pain. Neuropathic pain symptoms as identified with the mPDQ have been found to correlate with signs of central sensitisation in OA, as identified with QST.

SECONDARY OUTCOMES:
Premorbid IQ | Conducted once, at assessment visit approximately 10-15 minutes
  The National Adult Reading Test (NART) will serve as a measure of general premorbid IQ.
Depression/Anxiety | Conducted once, at assessment visit approximately 5-10 minutes
  The Hospital Anxiety and Depression Scale (HADS), a 14-item measure designed to assess anxiety and depression symptoms will be also used.
Sleep Quality: PSQI | Conducted once, at assessment visit approximately 5-10 minutes
  Sleep disturbances are common within people experiencing chronic pain and are associated with impaired cognitive function both in males and females. For that reason, the Pittsburgh sleep quality index (PSQI) will be utilised to assess sleeping patterns in people with chronic pain.
Physical function | Conducted once, at assessment visit approximately 6 minutes
  Functionality testing will be done using the 'time up and go' (TUG) test.
Physical function | Conducted once, at assessment visit approximately 5 minutes
  Functionality testing will be done using the 30-second sit to stand test (30CST)
Altruism/Decision making | Conducted once, at assessment visit approximately 5-10 minutes
  Participants will also complete a Dictator Game (DG) to explore the role of altruism in motivating subjects' behaviour in two independent settings, whereby participants will be given money (£10) and can donate some, all or none to: 1. an anonymous participant (75) and 2. a charity organisation.
Body mass index (BMI) | Conducted once, at assessment visit approximately 5 minutes
  Clinical assessment of body weight and height to determine BMI.
Inflammatory biomarkers | Conducted once, at assessment visit approximately 5-15 minutes for blood collection.
  Blood samples will be collected and serum sent for laboratory analysis to determine inflammatory biomarkers using RNA tubes.
biomarkers of insulin resistance | Once pre-assessment visit Urine sample will be collected at home and handed in at attendance of the visit 5 minutes
  Urine samples will be collected and sent for laboratory analysis to determine biomarkers of insulin resistance
gut microbiome measures. | Once post-assessment visit Faecal samples will be done home and sent back in prepaid envelope. 15 minutes
  Faecal (optional) samples will be collected and sent for laboratory analysis to determine gut microbiome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Valdes, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided